CLINICAL TRIAL: NCT03586570
Title: A Single-center, Double-blind, Placebo-controlled, Randomized Study to Investigate the Tolerability, Safety, and Pharmacokinetics After Multiple-dose Administration of 25 mg Aprocitentan in Healthy Japanese and Caucasian Subjects
Brief Title: A Study to Evaluate How Aprocitentan is Safe and How it is Absorbed and Broken Down in the Body of Japanese and Caucasian Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Collaborators: Janssen Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: ID-080-107
Record Dates: First submitted 2018-07-02; First posted 2018-07-13 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — aprocitentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Aprocitentan (Experimental)
  Interventions: Drug: Aprocitentan 25mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aprocitentan 25mg — Oral tablets in strength of 25 mg
  Arms: Aprocitentan
Drug: Placebo — Oral tablets matching aprocitentan tablets
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the tolerability, safety, and pharmacokinetics after multiple-dose administration of aprocitentan (25 mg) in healthy Japanese and Caucasian subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be of Caucasian or Japanese ethnicity
* Signed informed consent in a language understandable to the subject prior to any study-mandated procedure
* Body mass index (BMI) of 18.0 to 28.0 kg/m2 (inclusive) at Screening
* Systolic blood pressure 100-145 mmHg, diastolic blood pressure 50-90 mmHg, and pulse rate 45-90 bpm (inclusive), measured on the same arm, after 5 min in the supine position at Screening
* A woman of childbearing potential is eligible only if the following applies:

Negative serum pregnancy test at Screening,

Negative urine pregnancy test on Day -1,

Agreement to consistently and correctly use a reliable method of contraception from Screening up to at least 30 days after last study treatment administration

Japanese subjects only

* Subjects must be of native Japanese descent (all parents/grandparents of Japanese descent).
* Subjects must not have been away from Japan for more than 10 years (at Screening visit).
* Subject's lifestyle should not have changed significantly since relocation from Japan

Exclusion Criteria:

* Previous exposure to aprocitentan and/or macitentan.
* Known hypersensitivity to aprocitentan or treatments of the same class, or any of the excipients
* Pregnant or lactating women
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2018-09-10 (Actual)

PRIMARY OUTCOMES:
Cmax during the first and last dosing interval | From study treatment administration to 216 hours after last administration
Time to reach Cmax (tmax) during the first and last dosing interval | From study treatment administration to 216 hours after last administration
AUCτ on the first and last day of study treatment intake | From study treatment administration to 216 hours after last administration

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (1):
- Anaheim Clinical Trials, Anaheim, California, United States